CLINICAL TRIAL: NCT03782168
Title: Plasma Concentration of Biological Markers in Placental Abruption
Status: Terminated | Type: Observational
Why Stopped: IRB approval expired; failure to submit continuing review in time. Will re-open once IRB approval is reinstated.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 228485
Record Dates: First submitted 2018-12-10; First posted 2018-12-20 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2021-10

CONDITIONS: Abruptio Placentae
MeSH Terms: conditions — Abruptio Placentae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood for serum biomarkers and placental micro-particles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Placental Abruption: Mother-infant dyads with suspected or confirmed diagnosis of placental abruption
  Interventions: Other: There is no other intervention, only clinical treatment.
- Phenotypically-matched controlled group: Healthy mother-infant dyads admitted for delivery
  Interventions: Other: There is no other intervention, only clinical treatment.

INTERVENTIONS:
Other: There is no other intervention, only clinical treatment. — The purpose of this study is to determine how well maternal serum biomarkers and placental micro-particles (MP) correlate with PA. The sensitivity and specificity of these proteins will be analyzed to further increase our understanding of the pathological mechanisms involved in PA.

SUMMARY:
This will be a prospective study conducted on women with a suspected/confirmed diagnosis of placental abruption. Maternal blood samples will be taken at various points during the peripartum period. A healthy group of women admitted for delivery will act as a matched control and will have their blood sampled at similar time points. The primary outcome variables will include the total number of micro-particles, the number of micro-particles from each cell line (platelet, placental, endothelial etc.), and protein markers (specifically; placental growth factor (PlGF), soluble fms-like tyrosine kinase-1 (sFLT-1), vascular endothelial growth factor (VEGF), soluble endoglin (sEng)). Secondary outcomes if will examine the correlation between placental micro-particles, biomarkers, and extent of placental abruption.

DETAILED DESCRIPTION:
The purpose of this study is to determine how well maternal serum biomarkers and placental micro-particles (MP) correlate with PA. The sensitivity and specificity of these proteins will be analyzed to further increase our understanding of the pathological mechanisms involved in PA. The knowledge gained from this study has the potential to develop a diagnostic test for PA with the ability to improve outcomes for mother and baby through earlier diagnosis and targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - to 45-years old, inclusive
* Suspected or confirmed PA or phenotypically matched controls
* All modes of delivery
* Gestational age greater than 28 weeks
* Singleton pregnancy

Exclusion Criteria:

* Intrauterine fetal demise,
* Severe fetal anomalies (infant not expected to survive)
* Inability to communicate in English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mother-infant dyads with suspected or confirmed diagnosis of placental abruption and healthy mother-infant dyads admitted for delivery.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Determine the level of placental-derived MPs (Microparticles/mL) | Up to 75 minutes
  Determine quantitatively the level of placental-derived MPs which may be altered in 10 subjects with PA compared to 10 matched control subjects.
Identify biomarkers (picogram/mL) specifically, placental growth factor (PlGF), vascular endothelial growth factor (VEGF), soluble fms-like tyrosine kinase-1 (sFLT-1), and soluble endoglin (sEng) | Up to 75 minutes
  Determine quantitatively the level of biomarkers which may be altered in 10 subjects with PA compared to 10 matched control subjects.

SECONDARY OUTCOMES:
Examine the correlation between maternal serum total placental MPs and biomarkers to clinical symptomology and the severity of placental abruption after delivery. | Up to 75 minutes
  In order to evaluate the secondary outcome, the correlation between maternal serum total placental MPs, biomarkers to clinical symptomology, and the severity of placental abruption after delivery will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Shawrawi, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No